CLINICAL TRIAL: NCT02088580
Title: Feasibility and Tolerability of Adjunct Chronotherapy in Depressed Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chronotherapy Pilot
Record Dates: First submitted 2014-02-18; First posted 2014-03-17 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2013-09

CONDITIONS: Non-Psychotic Unipolar Depression; Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple Chronotherapy (Experimental): Total sleep deprivation, Sleep phase advance, and Bright light therapy.
  Interventions: Procedure: Triple Chronotherapy

INTERVENTIONS:
Procedure: Triple Chronotherapy
  Other Names: Sleep deprivation, Sleep phase advance, and Bright light therapy.

SUMMARY:
This study will attempt to study the effect of adjunctive chronotherapy (wake therapy, sleep phase advance, and bright light therapy) on acutely depressed inpatients. The investigators will attempt to recruit individuals admitted to the acute inpatient unit and study the results of the treatment on depressive symptoms, and suicidality.

DETAILED DESCRIPTION:
Acute depression, and suicidality continue to be significant causes of morbidity and mortality, and frequently result in acute inpatient hospitalization. Currently available treatments for depression have limitations for acute care including, either a slow onset of action such as is the case of pharmacotherapy, or high cost and limited availability such as is the case for ECT. This is exacerbated by ever shortening hospitalization times. Subsequently many of the individuals who are admitted for depression are discharged weeks before it can be expected for them to have symptomatic relief. Further more, in many cases treatment results in the trial of multiple medications before an effective treatment regimen is found (if such a treatment is found at all) (Rush, Trivedi et al. 2006). There is subsequently a great need for effective anti-depressant therapies with rapid onset of action, widespread availability, and cost effectiveness.

There is a consistent and expanding body of literature showing that chronotherapy is an effective, and rapid treatment of acute depression(Wu, Kelsoe et al. 2009, Martiny, Refsgaard et al. 2012, Echizenya, Suda et al. 2013). Published studies report response and remission rates in the range of 41-61%, 24-59% respectively acutely. Chronotherapy is a brief protocol that involves the combination of wake therapy (total sleep deprivation), sleep phase advance (a shift to an earlier sleep schedule with gradual normalization), and bright light therapy. The currently published reports have demonstrated efficacy in both unipolar and bipolar depression, and there has been reported stability of results for as long as 9 weeks (which was the longest designed study). Studies have been completed in real world clinical populations, which have included co-morbid populations, with the only groups showing a worsening of effect being those with psychotic depression (Benedetti, Zanardi et al. 1999), and those with panic disorder(Roy-Byrne, Uhde et al. 1986). The treatment itself has been well tolerated with a high percentage of individuals completing the procedure.

The current body of literature is encouraging, and the technique is being utilized clinically in some facilities (including our own institution), however there are still relatively few clinical trials published, and still unanswered questions that limit widespread clinical utility. One such issue is related to the high percentage of published trials performed outside of the US (although some have been done in the US). Because a high percentage of the studies have been done in other countries it is not clear if this procedure will translate well into the treatment paradigm in the US. Currently in the US, inpatient admission is restricted to individuals with severe, often highly treatment resistant disease that includes acute suicidality. To this writers knowledge there have not been any studies that specifically address suicidality. It is also not clear if patients in the US will tolerate the procedure. Tolerability has been addressed in many of the published papers, and in general the procedure is tolerated well with few if any side effects, however, again it is unclear how the procedure would be tolerated in clinical patients in the US.

ELIGIBILITY:
Inclusion Criteria:

* A current episode of non-psychotic major depression.
* Currently hospitalized.
* Age greater than 18.
* If bipolar illness, must not be a mixed state, and must be on a therapeutic dose of a mood stabilizer.

Exclusion Criteria:

* Urine drug screen positive for cocaine, or current alcohol abuse/dependence that requires detox.
* Current psychosis.
* Panic disorder.
* A history of seizures, uncontrolled severe headaches, stroke, or other neurologic illness that produces either gait abnormalities or a lowered seizure threshold.
* Medical illness that would make wake therapy intolerable, or significant cardiac disease.
* Cataracts, glaucoma, or other intrinsic eye condition.
* Currently taking light sensitizing medications.
* Current pregnancy which is routinely tested for prior to admission.
* Mental retardation, or dementia.
* Untreated sleep disorder such as Obstructive sleep apnea, narcolepsy, or PLMD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Day prior to total sleep deprivation, and then again over the next 4 consecutive days.
  Change Score of Pre and Post Hamilton depression depression scores
Columbia Suicide Severity Rating Scale | Daily throughout the treatment (Days 0-4)
  Change score in Columbia Suicide Severity Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States